CLINICAL TRIAL: NCT01226914
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Comparing Wound Drainage and Post-operative Complications With and Without the Use of EVICEL™ Fibrin Sealant in Thyroidectomy
Brief Title: A Trial Comparing Wound Drainage and Post-operative Complications With and Without the Use of EVICEL™ Fibrin Sealant in Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Shaun A. Nguyen, Associate Professor - Director of Clinical Research, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EVICEL
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Thyroid Neoplasm; Goiter
Keywords: EVICEL, Fibrin Sealant, Thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms; Goiter

STUDY DESIGN:
Intervention Model Description: prospective randomized placebo-controlled double-blind trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): For subjects in the placebo group, saline was drawn into the applicator and aerosolized in a similar fashion; it was allowed to remain in the wound during closure.
  Interventions: Drug: EVICEL
- Evicel (Experimental): For subjects in the treatment group, Evicel was applied in the usual manner by study personnel, with 5mL of each component drawn into a two-barrel syringe device and aerosolized using a pedal-controlled inert gas supply.
  Interventions: Drug: EVICEL

INTERVENTIONS:
Drug: EVICEL — EVICEL

SUMMARY:
Primary Objectives

* To compare the amount of post-operative wound drainage between the group of patients in which EVICEL™ spray is utilized (Arm A), and the group of patients in which an EVICEL™ placebo is utilized (Arm B).
* To compare the length of time to drain removal between Arm A and Arm B. Secondary objectives
* To compare the incident or rates of seroma, hematoma, and post-operative edema between the two groups.
* To compare the reported pain experienced in each group at selected time points using a standard numerical rating scale (NRS).
* To compare the length of hospital stay between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria

* Patients must have an initial diagnosis of thyroid neoplasmcarcinoma or goiter that requires total or hemithyroidectomy.
* Patients must have an ECOG performance status of 0-2
* Laboratory values must be within the following ranges:

  * Platelet count > 100 k/mm3
  * Hemoglobin > 10.0 g/dL
  * WBCs > 3.0 k/mm3
  * Total bilirubin < 2.6
  * Serum Creatinine < 2.0
  * PTT and PT/INR within institutional normal limits
* Patients must sign informed consent for study participation

Exclusion Criteria

* Evidence of distant metastasis of thyroid carcinoma
* Recurrent thyroid cancer
* Prior thyroid surgery or surgery to the neck.
* Patients with diagnosed coagulation disorders
* Prior irradiation to the neck area
* Prior chemotherapy for the current diagnosis
* Patients on therapeutic warfarin
* Patients with psychological or cognitive issues that, in the opinion of the investigator, will make them unable to adequately report pain levels
* Patients in an immune deficient state

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hornig, MD, Principal Investigator — Medical University of South Carolina; Shaun A Nguyen, M.D.,CPI, Study Director — Medical University of South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects undergoing total or partial thyroidectomy will be consented for this industry-sponsored prospective randomized placebo-controlled double-blind trial.
Pre-assignment Details: Subjects will be randomized to placebo or Evicel group based on a computer-generated random number sequence.
Period: Overall Study
Arm/Group | EVICEL Group | Placebo Group
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EVICEL Group: For subjects in the treatment group, Evicel was applied in the usual manner by study personnel, with 5mL of each component drawn into a two-barrel syringe device and aerosolized using a pedal-controlled inert gas supply.
- Placebo Group: For subjects in the placebo group, saline was drawn into the applicator and aerosolized in a similar fashion; it was allowed to remain in the wound during closure.
- Total: Total of all reporting groups
Arm/Group | EVICEL Group | Placebo Group | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (15.2) | 51.9 (11.5) | 50.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Amount of Post-operative Wound Drainage Between the Group of Patients in Which EVICEL™ Spray is Utilized (Arm A), and the Group of Patients in Which an EVICEL™ Placebo is Utilized (Arm B).
Description: First 8 hours output (mL), Total output (mL), Drain time (hours), Hospital stay (hours), AEs
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | EVICEL Group | Placebo Group
Number analyzed (Participants) | 28 | 27
mL | 96.3 [73.3 to 139.3] | 120 [68.8 to 161.5]

ADVERSE EVENTS:
Time Frame: Time from end of surgery to discharge was recorded for analysis. Adverse events were followed up to six months.
Arm/Group | EVICEL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 9/28 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVICEL (N=28) | Placebo (N=27)
hypocalcemia (Endocrine disorders) | 1 (1) | 2 (2)
hypocalcemia tetany (Endocrine disorders) | 2 (2) | 0 (0)
TVC paralysis (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Laryngeal edema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
asymptomatic hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-admit ED Incisional and Facial Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No